CLINICAL TRIAL: NCT01122329
Title: A Single-site Positron Emission Tomography (PET) Study of the Cerebral Metabolic Effects of AC-1202 (Axona®) Treatment in Mild-to-Moderate Alzheimer's Disease (AD)
Brief Title: A Positron Emission Tomography (PET) Study Evaluating Brain Metabolism of a Medical Food in Alzheimer's Disease
Acronym: AD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: John Douglas French Foundation (Other)
Responsible Party: Principal Investigator, Joshua Grill, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GG-AC-1202
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer Disease
Keywords: dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — caprylidene; AC-1202

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inactive food packet (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Axona® (Active Comparator)
  Interventions: Dietary Supplement: caprylidene

INTERVENTIONS:
Dietary Supplement: caprylidene — Axona® is dosed as a 40g packet mixed into 8 oz of liquid (Ensure) for 45 days
  Other Names: Axona®, AC-1202
  Arms: Axona®
Dietary Supplement: Placebo
  Arms: inactive food packet

SUMMARY:
This study will examine the brain metabolic effects of AC-1202 (Axona®), a medical food for Alzheimer's disease. Subjects who meet entry criteria will undergo H215O positron emission tomography prior to and 90 minutes after consumption of Axona® at baseline and then again after 45 days of treatment. Cognitive testing will also be conducted at baseline and day 45.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD (NINDS-ADRDA criteria(32))
* Age 50 - 90 (inclusive)
* MMSE range: 10 to 28
* Participants may be taking medications for AD, provided that the dose of these medications has been stable for > 90 days
* Proficiency in English to be able to perform cognitive tests
* A caregiver must be available to monitor and administer treatment and to accompany the subject to every clinical visit.

Exclusion Criteria:

* Inability for any reason to undergo PET/CT scans
* Previous treatment with AC-1202
* Allergic to milk or soy
* Presence of neurodegenerative disease other than AD
* History of stroke or other injury that could result in cognitive impairment
* Psychiatric disorder
* Diabetes mellitus
* Recent (<90 days) changes to medications prescribed for cognitive reasons or with the potential to impact cognition
* Irritable bowel syndrome (IBS) or other gastrointestinal conditions that could interfere with treatment compliance
* Any factor deemed by the investigator to be likely to interfere with study conduction

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Regional cerebral blood flow (rCBF) | At baseline
Regional cerebral blood flow (rCBF) | 90 minutes after initation of treatment with Axona®
Regional cerebral blood flow (rCBF) | 45 days after initation of treatment with Axona®

SECONDARY OUTCOMES:
Examine differences between ApoE ε4 carriers and noncarriers in changes on rCBF and cognition | At baseline
To examine the effect of AC-1202 on cognition | At baseline
Examine differences between ApoE ε4 carriers and noncarriers in changes on rCBF and cognition | At 90 minutes after initiation of treatment with Axona®
Examine differences between ApoE ε4 carriers and noncarriers in changes on rCBF and cognition | 45 days after initiation of treatment with Axona®
To examine the effect of AC-1202 on cognition | At 90 minutes after initiation of treatment with Axona®
To examine the effect of AC-1202 on cognition | 45 days after initiation of treatment with Axona®

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Grill, PhD, Principal Investigator — Mary S. Easton Center for Alzheimer's Disease Research at UCLA; John Ringman, MD, Study Chair — Mary S. Easton Center for Alzheimer's Disease Research at UCLA; Maryam Beigi, MD, Study Chair — Mary S. Easton Center for Alzheimer's Disease Research at UCLA; Ellen Woo, PhD, Study Chair — Mary S. Easton Center for Alzheimer's Disease Research at UCLA; Dan Silverman, MD, PhD, Study Chair — UCLA Department of Molecular and Medical Pharmacology; Cathy Lee, PhD, Study Chair — Mary S. Easton Center for Alzheimer's Disease Research at UCLA; Jeffrey Cummings, MD, Study Chair — Mary S. Easton Center for Alzheimer's Disease Research at UCLA
Locations (2):
- United States (2):
  - 200 Medical Plaza, UCLA Medical Center, Los Angeles, California
  - Center for Neurotherapeutics at UCLA, Los Angeles, California